CLINICAL TRIAL: NCT03102853
Title: Effects of a Healthy Nordic Diet on Abdominal Obesity, Body Weight Maintenance and Cardiometabolic Risk: a 2-year Randomised Controlled Study
Brief Title: Healthy Nordic Foods to Prevent Cardiometabolic Risk in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Lund University Hospital (Other)
Responsible Party: Principal Investigator, LieseLotte Cloetens, Principal Investigator, Lund University
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: NOVI377
Record Dates: First submitted 2017-03-22; First posted 2017-04-06 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Obesity; Cardiovascular Risk Factor; Diet Modification
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic diet (Active Comparator)
  Interventions: Other: Nordic diet
- Control diet (Other)
  Interventions: Other: Control diet

INTERVENTIONS:
Other: Nordic diet
  Arms: Nordic diet
Other: Control diet
  Arms: Control diet

SUMMARY:
This project will examine whether long-term consumption of healthy Nordic foods can maintain a healthy weight also after weight loss, and decrease abdominal fat accumulation and cardiometabolic risk. The study will be performed with the aim to achieve a substantial body weight loss in the first phase by prescribing a standardized low caloric dietary formula. The follow-up phase will be a body weight-maintenance period and the subjects will be randomised to a healthy Nordic diet group and a control diet group. During the study body weight will be monitored and other measurements will include insulin sensitivity, blood lipids and inflammation markers.

ELIGIBILITY:
Inclusion Criteria:

* age 25-67 years, BMI 30-40 kg/m2, waist circumference men >102cm and women > 88cm or sagittal abdominal diameter men >22cm and women >20cm, stable body weight

Exclusion Criteria:

* glucose >7.0 mmol/l, B-Hb1aC >48 mmol/L, triglycerides >4 mmol/l, total cholesterol >8 mmol/l, bloodpressure >160/100 mmHg, chronic disease, gastro-intestinal disease, hyper-/hypothyroidism, alcohol abuse, cancer, gastric bypass operation, gluten allergy, lactose intolerance, pregnancy

Ages: 25 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in sagittal abdominal diameter | Change from baseline to month 6, 12, 18, 24
Change in body weight | Change from baseline to month 6, 12, 18, 24

SECONDARY OUTCOMES:
Insulin sensitivity (HOMA-IR) | Before and after body weight loss/maintenance: baseline (week -6), 0 (after 6-week weight loss period, month 6, 12, 18, 24
Body fat and body lean mass (BIA) | Before and after body weight loss/maintenance: baseline (week -6), 0 (after 6-week weight loss period, month 6, 12, 18, 24
Blood lipids | Before and after body weight loss/maintenance: baseline (week -6), 0 (after 6-week weight loss period, month 6, 12, 18, 24
Blood pressure | Before and after body weight loss/maintenance: baseline (week -6), 0 (after 6-week weight loss period, month 6, 12, 18, 24
Markers of kidney and liver function | Before and after body weight loss/maintenance: baseline (week -6), 0 (after 6-week weight loss period, month 6, 12, 18, 24
Markers of inflammation and endothelial function | Before and after body weight loss/maintenance: baseline (week -6), 0 (after 6-week weight loss period, month 6, 12, 18, 24

CONTACTS AND LOCATIONS:
Locations (1):
- Biomedical Nutrition, Lund University and Unit for Diabetesstudies, Lund University Hospital, Lund, Sweden